CLINICAL TRIAL: NCT04760834
Title: Concussion in French Amateur Rugby: Descriptive Cross-sectional Survey About the Management and Knowledge of Players Over the 2019/2021 Seasons
Brief Title: Concussion in French Amateur Rugby : Survey About the Management and Knowledge of Players
Acronym: RUGBY-COM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/10
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Concussion
Keywords: Cerebral Concussion; Systems thinking; Injury management; Sport-related injury; Rugby union; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Complete a questionnaire to look for signs of concussion in the past. The questions also seek to collect data on participants' knowledge, concussion management and potential confounding factors

SUMMARY:
Rugby is a popular contact sport in France the majority of whom are amateur players. Concussion is one of the main risks given its potential severity and frequency (between 2.78 and 10 per 1,000 player hours). Faced with a concussion, stop sport activity, medical evaluation and a progressive resumption of activity are simple things to do to avoid an over-risk of injury and better recovery of the player. For this purpose, the rugby federation implement the blue card and the concussion declaration by clubs. A recent study showed that the directives of the federation are not sufficiently respected. The non-declaration problem is added knowing that around 50% of concussions are not declared. In professional rugby, the presence of a medical staff makes possible to optimize care as much as possible. In the amateur world, there are not always medical or paramedical personnel trained for this problem at the edge of the field when all the participants (player, coach, coaching) lack of knowledge on the subject and that the general practicer remains the referent for the concussion management. We will reach a dozen amateur rugby club to complete a questionnaire about concussions and conduct un formation session about this issue.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years of age or older
* Amateur rugby players in a club of New Aquitaine region who agreed to participate
* Licensed with the federation for 2019/2020 or 2020/2021 season
* Between the federal 1 and the 4th series

Exclusion Criteria:

- Refusal to complete the questionnaire

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amateur rugby players
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-09-16 (Estimated); Study Completion 2022-09-16 (Estimated)

PRIMARY OUTCOMES:
Number of cessation of any sporting activity | Inclusion
  Number of cessation of any sporting activity following a concussion during rugby practice, expressed as a percentage (ratio of the reported number of stops from any post-concussion sports activity to the number of rugby players reporting at least one concussion over the season).

SECONDARY OUTCOMES:
Number of post-concussion medical examination | Inclusion
  Reported number of post-concussion medical examination
Number of resumption of sporting activity | Inclusion
  Reported number of resumption of sporting activity carried out gradually after an initial stop in post concussion
Number of "yes" to Players's knowledge on the definition of concussion | Inclusion
  Players's knowledge of the definition of concussion and its management

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Cassoudesalle, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No